CLINICAL TRIAL: NCT05849597
Title: Dexmedetomidinine in the Prevention of Postoperative Delirium in the Intensive Care Unit After Cardiac Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Novi Sad (Other)
Responsible Party: Principal Investigator, Mihaela Preveden, Research Assistant, University of Novi Sad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 612-1/1
Record Dates: First submitted 2023-04-26; First posted 2023-05-09 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Intensive Care Unit Delirium
Keywords: open heart surgery; sedation; dexmedetomidine; postoperative delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Experimental): Evaluate the effects of dexmedetomidine for sedation of patients in the intensive care unit after open heart surgery
  Interventions: Drug: Dexmedetomidine
- Propofol (Active Comparator): Compare the clinical outcomes of the experimental group with the standard of care, i.e. sedation with propofol
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — Upon arrival to the intensive care unit after open heart surgery, the patients will be sedated with continuous dexmedetomidine infusion in doses 0.2-0.7 mcg/kg/h.
  Arms: Dexmedetomidine
Drug: Propofol — Upon arrival to the intensive care unit after open heart surgery, the patients will be sedated with continuous propofol infusion in doses 1-2 mg/kg/h.
  Arms: Propofol

SUMMARY:
This is a prospective, randomized, single blinded, controlled clinical trial designed to compare the clinical effects of sedation with dexmedetomidine versus propofol in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
The study will include adult patients of both sexes scheduled for elective cardiac surgery with the use of cardiopulmonary bypass (including coronary artery bypass grafting, valve repair/replacement, and combined).

The patients included in the study will be randomized in 1:1 ratio using computer generated numbers into two groups. The first group of patients, upon arrival to the intensive care unit will be sedated with continuous dexmedetomidine infusion in doses 0.2-0.7 mcg/kg/h. Dexmedetomidine infusion will be discontinued before weaning from mechanical ventilation and extubation. The second group of patients, upon arrival to the intensive care unit will be sedated with continuous propofol infusion in doses 1-2 mg/kg/h. Propofol infusion will also be discontinued before weaning from mechanical ventilation and extubation.

Sedation level will be assessed using Richmond Agitation and Sedation Scale (RASS) every two hours. Postoperative analgesia will be managed according to protocol (opioid analgesics, non-steroid anti-inflammatory drugs, paracetamol), with pain level assessment using visual analog scale (0 - no pain; 10 - unbearable pain).

The following data will be registered: age, sex, body mass index (BMI), hemoglobin, heart rate, and LVEF. Among the postoperative parameters, the following will registered: duration of mechanical ventilation (in hours), extubation time, ICU and hospital length of stay (in days), postoperative hemoglobin, blood product transfusion rates, occurrence of atrial fibrillation and assessment of delirium. Assessment of delirium will be performed using the confusion assessment method for intensive care unit (CAM-ICU) every 12 hours during five postoperative days.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing open heart surgery with the use of cardiopulmonary bypass (including coronary artery bypass grafting, valve repair/replacement, and combined)
* left ventricular ejection fraction (LVEF) >40%.

Exclusion Criteria:

* preoperative atrial fibrillation
* previous history of interventionally treated arrhythmias
* second and third degree atrioventricular block
* bradycardia with heart rate ≤50/min
* pacemaker
* renal or hepatic insufficiency
* emergency procedures
* history of serious mental illness, delirium, and severe dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of postoperative delirium | 5 days
  Assessment of delirium will be performed using the confusion assessment method for intensive care unit (CAM-ICU) at any time in the first five days after surgery

SECONDARY OUTCOMES:
MV duration | 30 days
  Duration of mechanical ventilation
ICU length of stay | 30 days
  Total duration of stay in the intensive care unit
Hospital length of stay | 30 days
  Total duration of stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela Preveden, MD, Principal Investigator — Institute of Cardiovascular Diseases of Vojvodina
Locations (1):
- Institute of Cardiovascular Diseases of Vojvodina, Kamenitz, Serbia

IPD SHARING:
Plan to Share IPD: No